CLINICAL TRIAL: NCT07166107
Title: EVOLV-Rx VA: Evaluating Opportunities to Decrease Low-Value Prescribing in Community Living Centers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 23-132; 1I01HX003849 (NIH)
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Low-Value Care
Keywords: Nursing Homes; Inappropriate Prescribing

STUDY DESIGN:
Intervention Model Description: In Aim 2, the investigators will conduct a randomized hybrid type 2 effectiveness implementation study applying a stepped wedge design to compare the EVOLV-Rx intervention to usual care. In the stepped wedge design, each CLC serves as its own control rather than sites being allocated to distinct control and intervention arms. This will enable all participating CLCs to receive the intervention, as is the desire of the operational partners in VISN 4 and will enhance the power to detect differences in outcomes relative to a traditional cluster randomized design. The stepped wedge design also allows for a sequential rollout of the intervention at each CLC. (Aims 1 and 3 are qualitative, and do not involve any intervention model).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stepped Wedge (Experimental): As part of the Stepped Wedge design, each CLC serves as its own control rather than sites being allocated to distinct control and intervention arms. All sites will receive the intervention.
  Interventions: Other: EVOLV-Rx dashboard

INTERVENTIONS:
Other: EVOLV-Rx dashboard — Using the TheraDoc® platform, the investigators will deploy a custom-designed EVOLV-Rx dashboard that incorporates all 18 components of the EVOLV-Rx metric. [Within TheraDoc®, the dashboard will display an automated report in the form of a patient list that includes the names, locations, and specific LVP practices to which Veterans under their care are subject. Pharmacists will then query specific patients on the list as part of their required medication review. The dashboard will provide detailed clinical decision support by identifying the specific EVOLV-Rx LVP criteria met by each flagged medication and provide access to the patient's full medication list, problem list, and laboratory or testing data contained within VISTA.] Pharmacists may use the EVOLV-Rx dashboard to track Veterans' receipt of LVP practices and quickly document actions related to the intervention, such as patient and family caregiver engagement, deprescribing LVP practices, or any other medications discontinued.

SUMMARY:
The investigators developed EVOLV-Rx (Evaluating Opportunities to Decrease Low-Value Prescribing), a novel clinical support tool to detect 18 evidence-based and clinically useful low-value prescribing practices in older adults. The objective is to conduct a hybrid study to assess the effectiveness and implementation of an EVOLV-Rx-based intervention to reduce LVP among older Veterans who reside in CLCs in VISN 4.

In Aim 1, the investigators will conduct focus groups of VISN 4 CLC leaders, clinicians, Veterans, and family caregivers, where the investigators will characterize the patient, clinician, and CLC-level barriers to and facilitators of implementation; and identify and tailor strategies to optimize the intervention's adoption and implementation. In Aim 2, the investigators will conduct a hybrid type 2 effectiveness implementation trial to compare the intervention to usual care, using a stepped wedge design in five VISN 4 CLCs. The primary effectiveness outcome is the count of low-value prescribing practices per 100 Veterans. In Aim 3, the investigators will conduct an embedded process evaluation to study implementation processes, their impact on outcomes, and iteratively improve the implementation of the intervention. The investigators will also conduct semi-structured interviews of clinicians, Veterans, and family caregivers to characterize the appropriateness, feasibility, acceptability, and perceived effectiveness of the intervention and implementation strategies employed.

DETAILED DESCRIPTION:
Background: More than half of Veterans aged 65 years who reside in Community Living Centers (CLCs) are subject to low-value prescribing, placing them at increased risk of adverse drug events, hospitalization, and death. CLCs represent an ideal setting to safely reduce low-value prescribing; however, no intervention to broadly reduce low-value prescribing has been successfully integrated into routine care or implemented at scale across CLCs. In response, the investigators developed EVOLV-Rx (Evaluating Opportunities to Decrease Low-Value Prescribing), a novel clinical support tool to detect 18 evidence-based and clinically useful low-value prescribing practices in older adults per an expert Delphi panel and further informed by patient, caregiver, and clinician input.

Significance: The objective is to conduct a hybrid study to assess the effectiveness and implementation of an EVOLV-Rx-based intervention to reduce LVP among older Veterans who reside in CLCs in VISN 4. This study will support VA's evolution as a learning healthcare system and is aligned with VA's key strategic healthcare priority of becoming the most age-friendly healthcare system in the United States. It also aligns with two VA HSR topic areas of interest, including improving healthcare quality and value and long-term care and aging. Innovation & Impact: EVOLV-Rx is a novel tool to detect low-value prescribing. Its unique characteristics and automated application will enable pharmacists to provide detailed recommendations to clinicians to prioritize medications for deprescribing with high clinical impact and that may be acceptably deprescribed from the perspective of patients and caregivers. EVOLV-Rx represents a substantial departure from the status quo, and its use will enhance deprescribing in CLCs and overcome several previously described implementation barriers.

Specific Aims: 1) To finalize the adaptable elements of, and implementation playbook for, the EVOLV-Rx intervention to reduce low-value prescribing for older Veterans residing in CLCs, 2) To assess the effectiveness of the EVOLV-Rx intervention to reduce low-value prescribing, 3) To evaluate and iteratively improve the implementation of the EVOLV-Rx intervention.

Methodology: Using the Theradoc clinical support platform, the intervention is an electronic EVOLV-Rx dashboard used by pharmacists to provide deprescribing recommendations to clinicians to reduce LVP as part of each Veteran's required medication review. The intervention will be translated into clinical practice in VISN 4 CLCs using a playbook of core implementation strategies previously employed in VA and additional strategies determined by key shareholders to address specific implementation barriers identified as part of the study. In Aim 1, the investigators will conduct focus groups of VISN 4 CLC leaders, clinicians, Veterans, and family caregivers, where the investigators will characterize the patient, clinician, and CLC-level barriers to and facilitators of implementation; and identify and tailor strategies to optimize the intervention's adoption and implementation. In Aim 2, the investigators will conduct a hybrid type 2 effectiveness implementation trial to compare the intervention to usual care, using a stepped wedge design in five VISN 4 CLCs. The primary effectiveness outcome is the count of low-value prescribing practices per 100 Veterans. In Aim 3, the investigators will conduct an embedded process evaluation to study implementation processes, their impact on outcomes, and iteratively improve the implementation of the intervention. The investigators will also conduct semi-structured interviews of clinicians, Veterans, and family caregivers to characterize the appropriateness, feasibility, acceptability, and perceived effectiveness of the intervention and implementation strategies employed.

Next Steps/Implementation: Leveraging VA infrastructure, the commitment of the investigators' operational partners, and the deep expertise of the research team, this proposal will result in a scalable intervention and accompanying implementation playbook to reduce low-value prescribing among Veterans receiving care in CLCs. It will also inform its deployment as a national multi-site trial to further evaluate and optimize its implementation throughout VA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 65+ admitted to a participating VISN 4 CLC at the time of the required medication review.

Exclusion Criteria:

* Veterans receiving hospice care, as the discontinuation of medications in EVOLV-Rx (e.g., benzodiazepines) may result in undue discomfort.

During both the usual care and intervention period of the study, the study coordinator will query the EVOLV-Rx dashboard weekly.

* The coordinator will ensure the presence of inclusion/exclusion criteria via chart review and using the EVOLV-Rx dashboard, they will then flag the patient if they are receiving hospice care and should be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1161 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Count of Low-Value Practices per 100 Veterans as per the EVOLV-rx metric | Baseline (starting an average of one year prior to implementation of intervention) through study completion, average time frame of 3.25 years of observation
  The primary effectiveness outcome is the count of LVP practices per 100 Veterans as per the EVOLV-Rx metric, which the investigators will consistently assess monthly from the start of the pre-implementation usual care phase through quarter 10. Data on LVP will be obtained from the VA Corporate Data Warehouse (CDW), including BCMA data, to fully capture Veterans' duration of medication use and pertinent diagnoses incorporated in the EVOLV-Rx criteria. A low-value medication will be characterized as discontinued if its discontinuation is sustained for 7 days, as this duration is unlikely to represent a temporary discontinuation of the medication. As per RE-AIM, maintenance will be determined via the assessment of the primary effectiveness outcomes at 6 and 12 months after the start of the intervention in each step of CLCs.

SECONDARY OUTCOMES:
Average Count of Long-term medications | Baseline (starting an average of one year prior to implementation of intervention) through study completion, average time frame of 3.25 years of observation
  Meds used for 28+ days prior to or during CLC admission
Proportion of Veterans with Polypharmacy and hyperpolypharmacy | Baseline (starting an average of one year prior to implementation of intervention) through study completion, average time frame of 3.25 years of observation
  Polypharmacy (5+ drugs), Hyperpolypharmacy (10+ drugs)
Proportion of Veterans with Adverse drug reactions | Baseline (starting an average of one year prior to implementation of intervention) through study completion, average time frame of 3.25 years of observation
  All VA ED/hospital transfers will be evaluated quarterly for potential Adverse Drug Reactions (ADR) via the Naranjo algorithm, which will be applied via EHR review. The Naranjo algorithm is a 10-point questionnaire to determine whether a suspected ADR is due to a drug rather than other factors.
Proportion of Veterans with Adverse drug withdrawal events | Baseline (starting an average of one year prior to implementation of intervention) through study completion, average time frame of 3.25 years of observation
  The Naranjo algorithm may also be applied to assess for adverse drug withdrawal events occurring in the period after medication withdrawal.
Average Count of ED visits/hospitalizations | Baseline (starting an average of one year prior to implementation of intervention) through study completion, average time frame of 3.25 years of observation
  As CLC residents may be transferred to the Emergency Department (ED) or hospitalized at a non-VA facility, the investigators will query both CDW and Medicare Data available through VIREC to assess the count of ED visits and hospitalizations. Count and review of ED visits/hospitalizations will be assessed retrospectively, given the delay in the availability of Medicare data.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Radomski, MD MS, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (2):
- United States (2):
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No